CLINICAL TRIAL: NCT04650724
Title: Single Arm, Single Center, Open Label Clinical Trial of BCMA Autologous Chimeric Antigen Receptor T Cell Infusion in Patients With BCMA Positive Recurrent or Refractory Multiple Myeloma
Brief Title: Clinical Study of T Cell Infusion Targeting BCMA Chimeric Antigen Receptor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-CART-BCMA-001
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell infusion agent targeting BCMA chimeric antigen receptor (Experimental)
  Interventions: Drug: T cell infusion agent targeting BCMA chimeric antigen receptor

INTERVENTIONS:
Drug: T cell infusion agent targeting BCMA chimeric antigen receptor — Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.

SUMMARY:
Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner, which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.

BCMA is a specific surface protein of B lymphocytes, which plays an important role in the development, proliferation and differentiation of B cells. BCMA is highly expressed in malignant mm plasma cells and provides a large number of anti apoptotic signals, which makes bcam an ideal target in targeted immunotherapy. At present, a variety of immunotherapy strategies targeting BCMA are being carried out in laboratory and clinical practice, which have achieved encouraging therapeutic effects in multiple myeloma and effectively promoted the development of targeted immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who voluntarily participated in the study and signed written informed consent;

  2. The age of signing informed consent is 14-65 years old;

  3. Patients with multiple myeloma were diagnosed according to the IMWG diagnostic criteria;

  4. The expression of BCMA was confirmed by flow cytometry or immunohistochemistry;

  5. The expected survival time was > 12 weeks;

  6. The main researchers and attending physicians believe that there is no other feasible and effective alternative treatment, such as hematopoietic stem cell transplantation;

  7. Relapsed or refractory multiple myeloma (mm) A. At least one complete regimen including induction, consolidation and maintenance of proteasome inhibitors and / or immunomodulators was performed at least once, and the interval between the two regimens was more than 3 months; B. According to the criteria of IMWG, recurrence was considered; C. Refractory patients (disease progression during standard treatment; efficacy of proteasome inhibitor combined with immunomodulator less than PR; efficacy after autologous stem cell transplantation less than PR; disease progression within 6 months after transplantation; progression and recurrence within 1 year after initial treatment); D. Recurrence occurred after allogeneic SCT treatment;

  8. The main organ functions are sound, including: A. Renal function: serum creatinine clearance rate > 40 ml / min / 1.73 m2, adjusted according to age / gender standard; B. Alanine transferase (ALT) was less than 2 times the normal maximum value of the same age; C. Bilirubin < 2.0 mg / dl; D. Echocardiography or multi gated angiography (MUGA) showed left ventricular short axis shortening (LVSF) ≥ 28%, or left ventricular ejection fraction (LVEF) ≥ 45%;

  9. ECOG physical status (PS) ≤ 2;

  10. The pregnant test results of fertile female subjects within 48 hours before infusion were negative, and they were not in lactation period; all subjects with reproductive potential should take adequate contraceptive measures from the beginning of the study to one year after the end of the study.

Exclusion Criteria:

* 1. Pregnant or lactating female patients;

  2. Participate in another clinical trial within 4 weeks before enrollment (3 months in case of monoclonal antibody clinical trial) or intend to participate in another clinical trial during the whole study period;

  3. Other anti BCMA treatments have been used in the past;

  4. Uncontrolled active infection; for example, there is a known history of human immunodeficiency virus; active hepatitis B or hepatitis C infection; HBV-DNA detection exceeds normal, etc;

  5. There is grade 2-4 acute or systemic chronic GVHD or GVHD under treatment;

  6. Cns-3 disease progression, or the presence of central nervous system parenchymal lesions that may increase the central nervous system toxicity; patients with active central nervous system leukemia infiltration;

  7. The researchers think that they are not suitable to participate in this clinical trial due to various reasons.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of AE or SAE | Study drug infusion within 12 weeks
  Incidence of AE or SAE with grade 3 or above related to study drug within 12 weeks of study drug infusion
ORR | Within 12 weeks after infusion of study drug
  Objective to study the clinical objective remission rate within 12 weeks after drug infusion

CONTACTS AND LOCATIONS:
Locations (1):
- No.3, Qingchun East Road, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided